CLINICAL TRIAL: NCT07005180
Title: A Phase 2a Multicenter, Randomized, Double-blind, Placebo-controlled Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, of HBI-002, an Oral Low-dose Carbon Monoxide (CO) Liquid Drug Product, Administered Daily Over 14 Days in Subjects With Parkinson's Disease (PD)
Brief Title: Low-dose Carbon Monoxide (HBI-002) Trial to Evaluate Safety, Tolerability, PK, and Biomarkers in Parkinson's Disease
Acronym: LoCaMoTE-PD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hillhurst Biopharmaceuticals, Inc. (Industry)
Collaborators: The Parkinson Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBI-002-221
Record Dates: First submitted 2025-02-28; First posted 2025-06-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; HBI-002; low dose carbon monoxide
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose (Experimental)
  Interventions: Drug: HBI-002
- Low Dose (Experimental)
  Interventions: Drug: HBI-002
- Placebo (Placebo Comparator)
  Interventions: Drug: Vehicle (placebo)

INTERVENTIONS:
Drug: HBI-002 — Oral liquid containing carbon monoxide
  Arms: High Dose; Low Dose
Drug: Vehicle (placebo) — Vehicle control (placebo)
  Arms: Placebo

SUMMARY:
A phase 2a multicenter, randomized, double-blind, placebo-controlled multiple dose study to evaluate the safety, tolerability, pharmacokinetics, of HBI-002, an oral low-dose carbon monoxide (CO) liquid drug product, administered daily over 14 days in subjects with Parkinson's disease (PD).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria before being enrolled into the study:

1. Signed informed consent.
2. Male or female 40-80 years of age
3. Non-smoker for at least 5 years with smoking defined as the use of smoked products (e.g. tobacco, marijuana, vaping or other)
4. No smoking in the home (i.e. not living with a smoker)
5. Body weight between 60 kg and 110 kg (inclusive) and with BMI less than 30 kg/m2 at screening and baseline
6. Diagnosis of PD according to the Movement Disorder Society within 60 months of screening
7. Hoehn and Yahr stage ≤ 3
8. PD therapy: use of ≥100 mg TID levodopa or equivalent dose with additional carbidopa/levodopa or other antiparkinsonian medication (e.g. dopamine agonists [e.g., pramipexole, ropinirole, rotigotine] and monoamine oxidase inhibitors [e.g., selegiline or rasagiline]) for ≥30 days of stable dosing
9. Good clinical response to levodopa therapy in the Site Investigator's opinion
10. Negative pregnancy test for females of childbearing potential
11. Where appropriate, subjects must be willing to use a highly effective method of contraception for the duration of the study and for 45 days thereafter

    1. Male subjects, without a vasectomy, whose partner is of childbearing potential, must use a condom and be instructed that their female partner should use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptive, injectable progesterone, subdermal implant or a tubal ligation. Male subjects are prohibited from donating sperm for the duration of the study and 60 days following the end of study visit.
    2. Female subjects of childbearing potential (not surgically sterilized and less than one year post-menopausal) should use a medically accepted form of contraception such as an IUD, diaphragm with spermicide, oral contraceptive, injectable progesterone, subdermal implant or a tubal ligation, and be instructed that their male partners should use a condom, if not vasectomized.
12. Subjects must be healthy as defined by the following.

    1. liver function: alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2X ULN
    2. total bilirubin ≤ 1.5X ULN
    3. renal function: creatinine clearance within normal range as assessed by Cockcroft and Gault calculation
    4. carboxyhemoglobin level by venous blood gas ≤ 3.5%
    5. the absence of current clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure, pulse rate, and respiratory rate measurement, 12-lead ECG, and clinical laboratory tests (hematology and clinical chemistries), as determined by the Site Investigator.
    6. HbA1c < 6.5%
13. Subjects must have a study partner who can observe the subject for at least 4 hours after dosing at home (non-clinic days) in order to monitor for indications of CO toxicity.
14. Subjects should live within 100 miles driving distance (door to door) of the site/clinic due to the need to carry study drug and ship study drug between the site/clinic and subject's home. Exceptions to this may be considered with Sponsor approval if it can be assured that the subject can transport study drug from clinic to home within two hours.

Exclusion Criteria:

Subjects who meet any of the following criteria will be ineligible for participation in the study:

1. Clinical signs indicating a parkinsonian syndrome other than idiopathic PD, specifically:

   1. Atypical parkinsonism, including parkinsonism due to drugs, metabolic disorders, encephalitis, cerebrovascular disease, normal pressure hydrocephalus, or other neurodegenerative disease.
   2. Supranuclear gaze palsy
   3. Signs of dementia (MoCA < 22)
   4. History of repeated strokes with stepwise progression of parkinsonian features
   5. History of repeated head injury
   6. History of definite encephalitis
   7. Cerebellar signs
   8. Early severe autonomic involvement
   9. Babinski sign present
2. Dysphagia with liquids
3. History of exposure to or current treatment with neuroleptic drugs.
4. History of dementia
5. Oxygen saturation by transcutaneous measurement ≤ 95% confirmed on repeat assessment (any time prior to the first dose)
6. Clinically significant ECG abnormalities (prolonged QTc greater than normal range, arrhythmia detected, bradycardia <45 bpm, tachycardia >120 bpm, AV block [second or greater degree], bundle branch block) or vital sign abnormalities (systolic blood pressure lower than 90 or above 140 mm Hg, diastolic blood pressure lower than 50 or above 90 mm Hg, or heart rate less than 45 or above 100 bpm or arrhythmia), as determined by the Site Investigator.
7. Renal failure requiring renal replacement therapy
8. History of:

   1. Serious cardiovascular diseases

      * History of angina pectoris
      * History of myocardial infarction or cardiac failure (NYHA from II to IV), myocardial insufficiency, symptomatic congestive heart failure with a documented ejection fraction below 45%
      * History of serious cardiac arrhythmia other than stable atrial fibrillation
      * History of stroke or occlusive peripheral vascular disease, brain vasospasm
   2. Structural brain disease or cerebrovascular disease with clinical significance, including intracranial space-occupying lesion
   3. Severe uncontrolled arterial hypertension
   4. Severe pulmonary disease (asthma, COPD, other)
   5. Specific psychiatric disorders, including hallucinations, delusions, pathologic gambling, alcohol or substance abuse or dependence
   6. Type 1 or type 2 diabetes mellitus, impaired glucose tolerance, metabolic syndrome, maturity onset diabetes of the young, and gestational diabetes.
   7. Pulmonary infiltrate or pneumonia within 6 months before screening or acute infection within 14 days of screening
   8. Seizures / epilepsy
   9. Autoimmune disease requiring prescribed immunomodulatory therapy
9. Alcohol abuse or dependence within one year prior to screening or regular use of alcohol within six months prior to the screening visit (defined as more than 14 units of alcohol per week; 1 Unit = 150 mL wine, 360 mL beer or 45 mL of 40% alcohol)
10. History of drug abuse or dependence
11. Positive result on drug screen for THC, cocaine, opiates/opioids, and methamphetamine
12. History of cancer, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin more than 3 months prior
13. Subject on domiciliary oxygen
14. Positive HBsAg, aHCV, or aHIV
15. Positive SARS-CoV-2 test within 10 days prior to study drug treatment
16. Weight loss or gain of more than 5 kg within 3 months of screening
17. Febrile or infective illness within 10 days prior to study drug treatment
18. Moderate or more severe depression (Geriatric Depression Scale (GDS) ≥9)
19. Suicide attempt or suicidal ideation within five years (Columbia-Suicide Severity Rating Scale (C-SSRS) defined as answering yes to items 4 or 5 on the C-SSRS, or history of suicide attempt in previous 5 years, or, in the Investigator's opinion, at serious risk of suicide.
20. Positive pregnancy test or breast feeding for females
21. Treatment with an investigational drug or medical device within the longer of 60 days or ten half-lives of the investigational agent
22. Simultaneous participation or previous participation within 60 days before screening in another clinical drug or medical device study
23. Persisting anemia with hemoglobin <9 g/dL
24. Blood transfusion within 42 days prior to the first administration of study drug
25. Exposure to any live vaccine within 28 days prior to study drug administration
26. Syncope or other cause of loss of consciousness within the last 2 years
27. Unwilling or unable to respond to follow-up phone calls
28. Unwilling or unable to communicate with study site staff by telephone
29. Unwilling or unable to comply with the requirements of the protocol
30. Any coincident disease or condition that in the opinion of the Site Investigator will confound the assessment of HBI-002 safety or efficacy
31. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Site Investigator, would make the subject inappropriate for entry into the study
32. History of allergic reactions to any of the drug product excipients
33. Contraindications to a routine lumbar puncture

    1. History of thrombocytopenia (platelet count <100,000)
    2. History of coagulopathy (INR >1.3, PTT >ULN)
    3. Current use of warfarin or other anticoagulants, or clopidogrel (Plavix)
    4. History of lumbar surgery or severe spinal arthritis
    5. Infection at LP site (may be included once resolved)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent AEs related to HBI-002 compared to placebo. | From treatment to 30 days after the end of treatment

SECONDARY OUTCOMES:
Pharmacokinetics as measured by carboxyhemoglobin (COHb) levels | Days 1 and 14

IPD SHARING:
Plan to Share IPD: Undecided